CLINICAL TRIAL: NCT03346837
Title: A Randomized, Open-Label, Four-Cohort, Parallel Design Study to Evaluate the Effect of Itraconazole or Rifampin on the Single-Dose Pharmacokinetics of BMS-986205 in Normal Healthy Participants
Brief Title: A Study to Evaluate the Effect of 2 Drugs on the Pharmacokinetics of BMS-986205 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CA017-051
Record Dates: First submitted 2017-11-06; First posted 2017-11-17 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Malignancies Multiple
MeSH Terms: interventions — linrodostat; Itraconazole; Rifampin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Inhibition (Cohort 1) (Experimental): Single oral dose BMS-986205
  Interventions: Drug: BMS-986205
- Inhibition (Cohort 2) (Experimental): Daily oral itraconazole doses for 24 days; single oral dose BMS-986205 on day 4
  Interventions: Drug: BMS-986205; Drug: Itraconazole
- Induction (Cohort 3) (Experimental): Single oral dose BMS-986205
  Interventions: Drug: BMS-986205
- Induction (Cohort 4) (Experimental): Daily oral rifampin doses for21 days; single oral dose BMS-986205 on day 8
  Interventions: Drug: BMS-986205; Drug: Rifampin

INTERVENTIONS:
Drug: BMS-986205 — BMS-986205
Drug: Itraconazole — Oral solution
  Arms: Inhibition (Cohort 2)
Drug: Rifampin — Tablet
  Arms: Induction (Cohort 4)

SUMMARY:
Assess the effects of itraconazole and rifampin on the pharmacokinetics, safety, and tolerability of BMS-986205.

DETAILED DESCRIPTION:
A randomized, open-label, parallel design study in healthy participants to assess the effects of itraconazole and rifampin on the single-dose pharmacokinetics of BMS-986205. Safety and tolerability data to be collected and assessed as well.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 18.0 to 32.0 kg/m2, inclusive
* Must have normal renal function demonstrated by GFR, calculated by Chronic Kidney Disease Epidemiology Collaboration formula
* Women must not be of childbearing potential (cannot become pregnant)

Exclusion Criteria:

* Any significant acute or chronic medical illness
* History of glucose-6-phosphodiesterase (G6PD) deficiency
* Personal or family history of cytochrome b5 reductase deficiency

Other protocol defined inclusion / exclusion criteria could apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to 25 days
  Measured by plasma concentration
AUC from time zero to time of last quantifiable concentration (AUC(0-T)) | Up to 25 days
  Measured by plasma concentration
AUC from time zero extrapolated to infinite time (AUC(INF)) | Up to 25 days
  Measured by plasma concentration

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 25 days
  Safety and tolerability as measured by incidence of AEs
Incidence of Serious Adverse Events (SAEs) | Up to 76 days
  Safety and tolerability as measured by incidence of SAEs
Number of participants with electrocardiogram abnormalities | Up to 25 days
Number of participants with physical examination findings abnormalities | Up to 25 days
Number of participants with clinical laboratory abnormalities | Up to 25 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Briston-Myers Squibb
Locations (1):
- PPD, Austin, Texas, United States

REFERENCES:
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/pages/investigator_inquiry_form.aspx
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls